CLINICAL TRIAL: NCT03622203
Title: Outcome of CHAllenging lesioNs and Patients Treated With Polymer Free Drug-CoatEd Stent ("Biofreedom"): the CHANCE a Multicenter Study
Brief Title: Outcome of CHAllenging lesioNs and Patients Treated With Polymer Free Drug-CoatEd Stent
Acronym: CHANCE
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Fabrizio D'Ascenzo, Principal Investigator, A.O.U. Città della Salute e della Scienza
Other Study IDs: CHANCE
Record Dates: First submitted 2018-05-18; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Coronary Disease; Drug Eluting Stent; STEMI
MeSH Terms: conditions — Coronary Disease; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- Real life patients: Patients who are often offered a Biofreedom in real life, that is those with active cancer or needing major surgery or on OAT (Oral Anticoagulation)
  Interventions: Device: Biofreedom
- Difficult coronary lesions: Patients with bifurcation and multivessel disease, that is those with an increased risk of ST
  Interventions: Device: Biofreedom
- STEMI: Patients with STEMI
  Interventions: Device: Biofreedom

INTERVENTIONS:
Device: Biofreedom — Use of Biofreedom in real life patients

SUMMARY:
Length of DAT (Dual Antiplatelet therapy) represents one of the most challenging choices for interventional cardiologist.

Prolonged DAT reduces risk of subsequent MI (Myocardial Infarction) with an increase in major bleedings, consequently with a neutral effect on survival [1].

Recently a Polymer-free Drug-Coated coronary stent has been tested in a randomized controlled trial with only one month of DAT due to its peculiar features, with an increased efficacy compared to BMS (Bare Metal Stent) and with a not negligible risk of ST at one year (about 2%)[2,3].

The RCT despite its promising design (inclusion of high risk patients like those with previous bleeding or with severe renal disease) showed a major limitation, that is:

1. patients who are often offered a Biofreedom in real life, that is those with active cancer or needing major surgery or on OAT (Oral Anticoagulation)
2. and patients with bifurcation and multivessel disease, that is those with an increased risk of ST [4]
3. STEMI patients [5] were underrepresented (less than 30%). Consequently we performed this multicenter study to evaluate safety and efficacy of Biofreedom in real life patients.

POCE (a composite end point of death, myocardial infarction, target lesion revascularization) and DOCE (cardiac death, MI-TLR and TLR) will be the primary end points, while its single components will be the secondary ones along stent thrombosis and with bleedings (Barc classification).

At least 12 months The Leaders FREE (2) reported an incidence of MACE of 9.4% at one year in overall patients. If there is a true difference in favour of the experimental treatment of 1.2%, then 870 patients are required to be 80% sure that the upper limit of a one-sided 95% confidence interval (or equivalently a 90% two-sided confidence interval) will exclude a difference when compared to non selected patients of more than 2% [5]

All patients implanting Biofreedom with these prespecified analysis:

1. Clinical

   * Diabetic patients (both insulin and not insulin depenent)
   * Requiring oral anticoagulation
   * On active cancer (that is requiring chemio or radio-therapy and or surgery)
   * Requiring surgery
   * STEMI
2. Interventional

   * Bifurcation (both provisional both 2 stents)
   * Multivessel
   * Ostial

DETAILED DESCRIPTION:
Our interest is to test the performance of these stents in real life patients

ELIGIBILITY:
Inclusion Criteria:

1. Clinical

   * Diabetic patients (both insulin and not insulin depenent)
   * Requiring oral anticoagulation
   * On active cancer (that is requiring chemio or radio-therapy and or surgery)
   * Requiring surgery
   * STEMI
2. Interventional

   * Bifurcation (both provisional both 2 stents)
   * Multivessel
   * Ostial

Exclusion

1. clinical less than 18 years old or more than 80
2. interventional last remaing vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients implanting Biofreedom with these prespecified analysis:
  1. Clinical
     * Diabetic patients (both insulin and not insulin depenent)
     * Requiring oral anticoagulation
     * On active cancer (that is requiring chemio or radio-therapy and or surgery)
     * Requiring surgery
     * STEMI
  2. Interventional
     * Bifurcation (both provisional both 2 stents)
     * Multivessel
     * Ostial
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of POCE (primary patient-oriented endpoint) | At least 6 months
  Incidence of POCE (a composite and mutual exclusive end point of death, myocardial infarction, target lesion revascularization)

SECONDARY OUTCOMES:
Incidence of Death | At least 6 months
  Incidence of Death
Incidence of Myocardial Infarction | At least 6 months
  Incidence of Myocardial Infarction
Incidence of TLR | At least 6 months
  Incidence of target lesion revascularization
Incidence of Cardiac Death | At least 6 months
  Incidence of Cardiac Death
Incidence of MI-TLR | At least 6 months
  Incidence of Myocardia Infarction TLR

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio D'Ascenzo, Principal Investigator — Città della Salute e Della Scienza di Torino

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mauri L, Kereiakes DJ, Yeh RW, Driscoll-Shempp P, Cutlip DE, Steg PG, Normand SL, Braunwald E, Wiviott SD, Cohen DJ, Holmes DR Jr, Krucoff MW, Hermiller J, Dauerman HL, Simon DI, Kandzari DE, Garratt KN, Lee DP, Pow TK, Ver Lee P, Rinaldi MJ, Massaro JM; DAPT Study Investigators. Twelve or 30 months of dual antiplatelet therapy after drug-eluting stents. N Engl J Med. 2014 Dec 4;371(23):2155-66. doi: 10.1056/NEJMoa1409312. Epub 2014 Nov 16. PMID 25399658
- [Background] Urban P, Meredith IT, Abizaid A, Pocock SJ, Carrie D, Naber C, Lipiecki J, Richardt G, Iniguez A, Brunel P, Valdes-Chavarri M, Garot P, Talwar S, Berland J, Abdellaoui M, Eberli F, Oldroyd K, Zambahari R, Gregson J, Greene S, Stoll HP, Morice MC; LEADERS FREE Investigators. Polymer-free Drug-Coated Coronary Stents in Patients at High Bleeding Risk. N Engl J Med. 2015 Nov 19;373(21):2038-47. doi: 10.1056/NEJMoa1503943. Epub 2015 Oct 14. PMID 26466021
- [Background] Garot P, Morice MC, Tresukosol D, Pocock SJ, Meredith IT, Abizaid A, Carrie D, Naber C, Iniguez A, Talwar S, Menown IBA, Christiansen EH, Gregson J, Copt S, Hovasse T, Lurz P, Maillard L, Krackhardt F, Ong P, Byrne J, Redwood S, Windhovel U, Greene S, Stoll HP, Urban P; LEADERS FREE Investigators. 2-Year Outcomes of High Bleeding Risk Patients After Polymer-Free Drug-Coated Stents. J Am Coll Cardiol. 2017 Jan 17;69(2):162-171. doi: 10.1016/j.jacc.2016.10.009. Epub 2016 Oct 30. PMID 27806919
- [Background] D'Ascenzo F, Bollati M, Clementi F, Castagno D, Lagerqvist B, de la Torre Hernandez JM, ten Berg JM, Brodie BR, Urban P, Jensen LO, Sardi G, Waksman R, Lasala JM, Schulz S, Stone GW, Airoldi F, Colombo A, Lemesle G, Applegate RJ, Buonamici P, Kirtane AJ, Undas A, Sheiban I, Gaita F, Sangiorgi G, Modena MG, Frati G, Biondi-Zoccai G. Incidence and predictors of coronary stent thrombosis: evidence from an international collaborative meta-analysis including 30 studies, 221,066 patients, and 4276 thromboses. Int J Cardiol. 2013 Jul 31;167(2):575-84. doi: 10.1016/j.ijcard.2012.01.080. Epub 2012 Feb 22. PMID 22360945
- [Background] Naber CK, Urban P, Ong PJ, Valdes-Chavarri M, Abizaid AA, Pocock SJ, Fabbiocchi F, Dubois C, Copt S, Greene S, Morice MC; LEADERS FREE Investigators. Biolimus-A9 polymer-free coated stent in high bleeding risk patients with acute coronary syndrome: a Leaders Free ACS sub-study. Eur Heart J. 2017 Apr 1;38(13):961-969. doi: 10.1093/eurheartj/ehw203. PMID 27190095
- [Background] Blackwelder WC. "Proving the null hypothesis" in clinical trials. Control Clin Trials. 1982 Dec;3(4):345-53. doi: 10.1016/0197-2456(82)90024-1. PMID 7160191
- [Derived] Gallone G, D'Ascenzo F, Boccuzzi G, Cortese B, Di Biasi M, Omede P, Capodanno D, Cerrato E, Vicinelli P, Infantino V, Poli A, Ugo F, Conrotto F, Grigis G, Varbella F, Latini RA, D'Urbano M, Montabone A, Senatore G, Ferrara E, D'Amico M, De Ferrari GM, Ielasi A. Real-world reasons and outcomes for 1-month versus longer dual antiplatelet therapy strategies with a polymer-free BIOLIMUS A9-coated stent. Catheter Cardiovasc Interv. 2020 Sep 1;96(3):E248-E256. doi: 10.1002/ccd.28757. Epub 2020 Feb 3. PMID 32012453
- [Derived] D'Ascenzo F, Gallone G, Boccuzzi G, Cortese B, Di Biasi M, Capodanno D, Vicinelli P, Infantino V, Poli A, Grigis G, Varbella F, De Ferrari GM, Ielasi A; Collaborators. Dual antiplatelet therapy strategies and clinical outcomes in patients treated with polymer-free biolimus A9-coated stents. EuroIntervention. 2020 Feb 7;15(15):e1358-e1365. doi: 10.4244/EIJ-D-19-00450. PMID 31334704